CLINICAL TRIAL: NCT05284266
Title: Surgical Treatment of Lipedema in Norway - a National Multicenter Study
Brief Title: The National Lipedema Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haraldsplass Deaconess Hospital (Other)
Collaborators: St. Olavs Hospital (Other); University Hospital of North Norway (Other); Sykehuset Telemark (Other Government); University of Bergen (Other); Klinbeforsk (Other); Helse Vest (Other)
Responsible Party: Principal Investigator, Hildur Skuladottir, Medical Doctor, PhD, Haraldsplass Deaconess Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 239087
Record Dates: First submitted 2022-03-08; First posted 2022-03-17 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Lipedema
Keywords: Liposuction; Conservative treatment; Intermittent pneumatic compression; Lipoedema; Compression therapy; Self management; Dietary management
MeSH Terms: conditions — Lipedema

STUDY DESIGN:
Intervention Model Description: Eligible patients are randomized to two different conservative treatment protocols;either standard conservative treatment (SCT) or standard treatment plus additional lymphedema treatment (intermittent pneumatic compression -IPC). After 6 months the effects of the conservative treatment are evaluated. Patients who still want surgery and fulfill the criteria are randomized (1:1) to early (cases(liposuction initiated 6-9 months after inclusion)) or late surgery (controls (liposuction initiated 18-21 months after inclusion)). Randomization to the surgical group is stratified by conservative treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Standard conservative treatment (Active Comparator): Standard conservative treatment consisting of:
  * Physical therapy, including compression garment and exercise program
  * Self-care program
  * Individual counseling from a clinical dietician
  Interventions: Other: Standard conservative treatment
- Standard treatment plus additional lymphedema treatment (Experimental): Standard conservative treatment consisting of:
  * Physical therapy, including compression garment and exercise program
  * Self-care program
  * Individual counseling from a clinical dietician Additional lymphedema treatment consisting of intermittent pneumatic compression (IPC)
  Interventions: Other: Standard conservative treatment with Intermittent Pneumatic Compression (IPC)
- Surgical group: Liposuction (Experimental): Early liposuction, 6-9 months after inclusion in study.
  Interventions: Procedure: Liposuction early
- Surgical group: Control (Active Comparator): Late liposuction, 18-21 months after inclusion. This group functions as a control group for 1 year before enrolment in the Liposuction group.
  Interventions: Procedure: Liposuction late

INTERVENTIONS:
Procedure: Liposuction early — Liposuction 6-9 months after inclusion
  Arms: Surgical group: Liposuction
Procedure: Liposuction late — Liposuction 18-21 months after inclusion
  Arms: Surgical group: Control
Other: Standard conservative treatment — Standard Conservative treatment consisiting of:
  Physical therapy, including compression garment and exercise program, Self-care program
  Arms: Standard conservative treatment
Other: Standard conservative treatment with Intermittent Pneumatic Compression (IPC) — Physical therapy, including compression garment and exercise program, Self-care program and Intermittent Pneumatic Compression (IPC)
  Arms: Standard treatment plus additional lymphedema treatment

SUMMARY:
Lipedema is a chronic condition with a symmetrical accumulation of painful fatty tissue primarily affecting the limbs, sparing hands, feet and trunk. The subcutaneous fatty tissue is disproportionately voluminous and may have a different microstructure and metabolism than the patient's regular fatty tissue. The condition affects almost exclusively women and usually debuts around puberty. Lipedema seems to have a hereditary component, may be affected by hormonal variations and worsens with obesity. Guidelines advocate conservative treatment with compression therapy, weight management, physical activity, life style changes and psychological support;and in some cases surgical treatment such as bariatric surgery and liposuction.

Treatment of lipedema is indicated when the condition causes significant pain and inhibits the patient's everyday activities. Well-designed randomized controlled studies on lipedema are lacking.

The Ministry of Health and Care Services in Norway has found the scientific documentation for the effects of liposuction to be insufficient and has recommended that surgical treatment of lipedema should be evaluated through a 5-year clinical trial. A national task force, consisting of representatives from all four regional health authorities in Norway has been set up. This task force has now initiated this study. A national multi-center study with homogenous treatment protocols can provide globally sought insight on lipedema and the effect of its treatment regimes, and the findings will be important to adjust future treatment strategies regarding both effect and cost/effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* female
* age 20-65 years
* significant pain from lipedema
* lipedema stage 1-2 or localized stage 3

Exclusion Criteria:

* Non-fluency in the Norwegian language
* pregnancy
* current malignancy
* previous surgical treatment for lipedema
* smoking
* BMI > 28
* serious comorbidities such as cardiac-, pulmonary-, renal disease
* unwillingness to wear compression garments

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2022-03-11 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Effect of liposuction on lipedema pain | 12 months after the last liposuction surgery
  Assess the effect of liposuction on lipedema pain (Visual Analog Scale (VAS). VAS consists of a 10 cm line, with two end points representing 0 (no pain) and 10 (worst possible pain).

SECONDARY OUTCOMES:
Effect of liposuction on quality of life and everyday activities for patients with lipedema | 12 months after the last liposuction surgery
  Assess the effect of liposuction on quality of life and everyday activities (RAND-36)

OTHER OUTCOMES:
Effect of different conservative treatments on lipedema pain and quality of life and everyday activities for patients with lipedema | 6 months after inclusion
  Effect of two different conservative treatments strategies on pain and everyday activities (RAND-36)
Adverse effect of liposuction | 12 months after last liposuction surgery
  Assess possible adverse effects of liposuction
Effect of liposuction on the need for conservative treatment | 3 years after last liposuction surgery
  Assess whether having undergone liposuction changes the need for conservative treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hildur Skuladottir, PhD, Principal Investigator — Haraldsplass Deaconess Hospital
Locations (1):
- Haraldsplass Deaconess Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Yes
Data will be available after publication of outcomes.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be available after publication of outcomes.